CLINICAL TRIAL: NCT01208272
Title: A Randomized Comparison of Group-Behavioral Therapy and Group Interpersonal Psychotherapy for the Treatment of Overweight Individuals With Binge-Eating Disorder
Brief Title: Psychological Treatment of Overweight Binge Eaters
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Denise E. Wilfley, Ph.D., Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R29MH051384 (NIH)
Record Dates: First submitted 2010-08-31; First posted 2010-09-23 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Binge Eating Disorder; Cognitive Therapy/Methods; Mental Disorders/Epidemiology; Obesity/Epidemiology; Obesity/Therapy
Keywords: Body Mass Index; Bulimia/therapy; Comorbidity; Interpersonal Relations; Psychotherapy/methods
MeSH Terms: conditions — Binge-Eating Disorder; Mental Disorders; Obesity; Bulimia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- Binge Eating Disorder/Therapy (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT); Behavioral: Interpersonal Therapy (IPT)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT)
Behavioral: Interpersonal Therapy (IPT)

SUMMARY:
Cognitive-behavioral therapy (CBT) has documented efficacy for the treatment of binge eating disorder (BED). Interpersonal psychotherapy (IPT) has been shown to reduce binge eating but its long-term impact and time course on other BED-related symptoms remain largely unknown. This study compares the effects of group CBT and group IPT across BED-related symptoms among overweight individuals with BED.

DETAILED DESCRIPTION:
Cognitive-behavioral therapy (CBT) has documented efficacy for the treatment of binge eating disorder (BED). Interpersonal psychotherapy (IPT) has been shown to reduce binge eating but its long-term impact and time course on other BED-related symptoms remain largely unknown. This study compares the effects of group CBT and group IPT across BED-related symptoms among overweight individuals with BED. METHODS: One hundred sixty-two overweight patients meeting DSM-IV criteria for BED were randomly assigned to 20 weekly sessions of either group CBT or group IPT. Assessments of binge eating and associated eating disorder psychopathology, general psychological functioning, and weight occurred before treatment, at posttreatment, and at 4-month intervals up to 12 months following treatment. RESULTS: Binge-eating recovery rates were equivalent for CBT and IPT at posttreatment (64 [79%] of 81 vs 59 [73%] of 81) and at 1-year follow-up (48 [59%] of 81 vs 50 [62%] of 81). Binge eating increased slightly through follow-up but remained significantly below pretreatment levels. Across treatments, patients had similar significant reductions in associated eating disorders and psychiatric symptoms and maintenance of gains through follow-up. Dietary restraint decreased more quickly in CBT but IPT had equivalent levels by later follow-ups. Patients' relative weight decreased significantly but only slightly, with the greatest reduction among patients sustaining recovery from binge eating from posttreatment to 1-year follow-up. CONCLUSIONS: Group IPT is a viable alternative to group CBT for the treatment of overweight patients with BED. Although lacking a nonspecific control condition limits conclusions about treatment specificity, both treatments showed initial and long-term efficacy for the core and related symptoms of BED.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV research criteria for binge-eating disorder
* Average of greater than or equal to 2 days of binge eating per week for at least 6 months' duration
* Marked stress regarding binge eating
* At least 3 to 5 associated behavioral features (e.g. eating when not physically hungry) Other study criteria
* 18-65 years old
* Body mass index, 27-48 kg/m squared

Exclusion Criteria:

* Pregnant or planning to become pregnant
* Taking weight-affecting or psychotropic medications
* Psychiatric conditions warranting immediate treatment
* Current enrollment in psychotherapy or a weight loss program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 1994-04; Primary Completion 1998-03 (Actual); Study Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
To investigate the short and long-term efficacy of two treatments for binge eating among the overweight: Group Cognitive-Behavior (CBT) and Group Interpersonal Therapy (IPT).
  Assessments of binge eating and associated eating disorder paychopathology, general psychological functioning, and weight occurred before treatment, at post treatment, and at 4-month intervals up to 12 months following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Denise E Wilfley, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Yale University, New Haaven, Connecticut
  - Yale University, New Haven, Connecticut

REFERENCES:
- [Result] Wilfley DE, Welch RR, Stein RI, Spurrell EB, Cohen LR, Saelens BE, Dounchis JZ, Frank MA, Wiseman CV, Matt GE. A randomized comparison of group cognitive-behavioral therapy and group interpersonal psychotherapy for the treatment of overweight individuals with binge-eating disorder. Arch Gen Psychiatry. 2002 Aug;59(8):713-21. doi: 10.1001/archpsyc.59.8.713. PMID 12150647
- [Derived] Hilbert A, Bishop ME, Stein RI, Tanofsky-Kraff M, Swenson AK, Welch RR, Wilfley DE. Long-term efficacy of psychological treatments for binge eating disorder. Br J Psychiatry. 2012 Mar;200(3):232-7. doi: 10.1192/bjp.bp.110.089664. Epub 2012 Jan 26. PMID 22282429